CLINICAL TRIAL: NCT01321515
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Famciclovir Tablets Under Fasting Conditions
Brief Title: Bioequivalency Study of Famciclovir 500 mg Tablets Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Executive Director, Drug Regulatory and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FAMC-T500-PVFS-1
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Herpes
MeSH Terms: conditions — Herpes Simplex | interventions — Famciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: famciclovir — 500 mg tablet
  Other Names: FAMVIR

SUMMARY:
The objective of this study was to prove the bioequivalence of Famciclovir 500 mg Tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to famciclovir, penciclovir or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Benno G Roesch, M.D., Principal Investigator — Advanced Biomedical Research
Locations (1):
- Advanced Biomedical Research, Inc., Hackensack, New Jersey, United States